CLINICAL TRIAL: NCT06477796
Title: A Sleep Intervention to Improve Quality of Life and Symptom Management in Veterans With the Polytrauma Clinical Triad
Brief Title: Improving Sleep in Veterans With the Polytrauma Clinical Triad
Acronym: LIONv2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: D4822-R; I01RX004822 (NIH)
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Traumatic Brain Injury; Post-traumatic Stress Disorder; Chronic Pain
Keywords: polytrauma clinical triad; TBI; PTSD
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Chronic Pain | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive MBLT or a sham/no-light control. Subjects randomized to receive MBLT will be given a light box (LightPad, Aurora Light Solutions) to take home. Subjects randomized to receive the sham/no-light control will be given a modified negative ion generator.
Who Masked: Participant
Masking Description: Participants will be blinded to the intervention by way of study personnel's description. Subjects will be told that both devices may or may not be active and thus, will be unaware that all light boxes are active and all negative ion generators are inactivated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning Bright Light Therapy (Experimental): Morning bright light: Sitting in front of a lightbox for 60 minutes every morning within 120 minutes of waking up.
  Interventions: Device: Morning Bright Light Therapy
- Negative Ion Generator (Sham Comparator): Negative ion generator: Sitting in front of a modified negative ion generator for 60 min every morning within 120 minutes of waking up.
  Interventions: Device: Negative Ion Generator

INTERVENTIONS:
Device: Morning Bright Light Therapy — Morning bright light: Sitting in front of a lightbox for 60 minutes every morning within 120 minutes of waking up.
  Other Names: Lightbox, light therapy
  Arms: Morning Bright Light Therapy
Device: Negative Ion Generator — Negative ion generator: Sitting in front of a modified negative ion generator for 60 min every morning within 120 minutes of waking up.
  Arms: Negative Ion Generator

SUMMARY:
The "polytrauma clinical triad" (PCT), a highly disabling constellation of factors, is defined by the coexistence of traumatic brain injury, post-traumatic stress disorder, and chronic pain. Veterans with the PCT are medically complex, often refractory to conventional therapies, and suffer from additional related chronic sequela. Notably, sleep disturbances and cognitive impairment, which the investigators hypothesize are significant contributing factors to these functional impairments and an impediment toward rehabilitation. Thus, the investigators' research aims to intervene "at the level of sleep", and by improving sleep, improve these interconnected, disabling, and difficult to treat enduring complexities associated with the PCT - ultimately to improve Veteran quality of life, functional independence, and restorative function. The investigators predict that the proposed intervention, morning bright light therapy, which is cost-effective, rapidly deployable and home-based, will be effective in improving sleep and overall PCT symptom management, thereby, resulting in a measurable and impactful improvement in quality of life.

DETAILED DESCRIPTION:
The co-existence of traumatic brain injury, post-traumatic stress disorder (PTSD), and chronic pain defines the clinical entity referred to as the "polytrauma clinical triad" (PCT). Well recognized to be highly prevalent and disabling in US military service members and Veterans, those with the PCT are traditionally viewed as the most disabled cases and most refractory to conventional therapies. Central to the challenge in effectively treating Veterans with the PCT is the bi-directional, mutually reinforcing relationship between these conditions. Further complicating is the influence of sleep and cognitive impairment, both of which are widely regarded as primary contributing chronic sequela associated with the PCT. The specific contribution from sleep in exacerbating this clinical picture is supported by extensive scientific precedent demonstrating impairments in sleep intensify and worsen these related sequela (e.g., cognitive impairment, pain management, and PTSD symptom severity), which in turn, contribute to further impairment in sleep. Accordingly, an effective intervention targeting sleep may alleviate rehabilitative pressure on these associated sequelae and facilitate breaking out of this vicious cycle (i.e., poor sleep exacerbating outcomes, and in turn, further impairing sleep).

Recent work from the investigators' laboratory demonstrate promise for a simple, at home, non-pharmacologic and cost-effective, sleep focused intervention: morning bright light therapy (MBLT). The investigators have demonstrated robust feasibility, acceptability, and limited efficacy for MBLT to improve sleep, and thereby, improve cognitive function, PCT symptom management and overall quality of life in this medically complex and vulnerable population. Accordingly, this proposal aims to extend the foundational work from the CDA-2 to inform a prospective phase II placebo-controlled randomized clinical trial examining effectiveness for MBLT as a sleep- based intervention in Veterans with the PCT.

Specific aims designed to test this hypothesis are to determine effectiveness for MBLT to improve 1) sleep, 2) cognition, and 3) PCT symptom management in Veterans with the PCT. The investigators propose to enroll n=138 Veterans, randomized 2:1 to MBLT (10,000 lux light exposure for 60 min within 120 min of waking for 4-weeks) or a no- light sham-MBLT condition (as previously published using the same duration/timing). Sleep, cognition and PCT symptom management will be assessed through a novel combination of subjective/self-report, objective measures, and ecological momentary assessment sampling. Specific objective assessments include wrist- based actigraphy and as exploratory outcome in a sub-set of participants, home-based overnight polysomnography. Outcomes will be assessed pre- and post-intervention, with follow-up at 6- and 12-weeks post-intervention.

It is expected the proposed work will demonstrate effectiveness for MBLT to improve sleep, cognition, and PCT symptom management including ameliorating chronic pain and improving quality of life, in Veterans with the PCT. This project will demonstrate, 1) an effective treatment option, alone or in combination with existing rehabilitative efforts, in Veterans with the PCT, and 2) sleep-wake disturbances may be implicated in the pathogenesis of these functional impairments, thereby establishing greater precedent for targeting sleep as a meaningful primary and/or adjunctive rehabilitative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* English speaking with phone and internet access
* Current self-reported sleep disturbances
* Clinical stable for current pharmacologic or behavioral health treatments for depression, anxiety, sleep and pain
* Documented history of TBI

Exclusion Criteria:

* Decisional impairment and/or dementia
* Current usage of a lightbox or negative ion generator
* Shift work
* History of macular degeneration and/or bipolar disorder
* Evidence for suicidal ideation
* Cancer diagnosis within the past 6 months
* Surgery within the past 6 months
* Substance abuse within the past 6-12 months
* Significant impairing post-stroke residual hemiparesis

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency via wrist based actigraphy | Pre- and post-4 weeks of MBLT or sham treatment
  Sleep efficiency is defined by the total time asleep divided by total time spent in bed

SECONDARY OUTCOMES:
Self-reported sleep quality via the Pittsburgh Sleep Quality Index | Pre- and post-4 weeks of MBLT or sham treatment
  The Pittsburgh Sleep Quality Index is a validated questionnaire assessing metrics related to sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan E Elliott, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No